CLINICAL TRIAL: NCT06149052
Title: Effects of SMART Training Intervention Versus Foot Intensive Rehabilitation (FIRE) on Strength and Performance in Athletes With Chronic Ankle Instability
Brief Title: Effects of SMART VS FIRE Training in Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCRS/1021 Wajeeha
Record Dates: First submitted 2023-08-18; First posted 2023-11-28 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Chronic Ankle Instability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: warm up exercises with SMART training (Active Comparator): For sensory stimulation planter massage was given, and it was applied to entire planter surface. Grade III anterior to posterior talocrural joint mobilization was given. For balance, single and double leg stance was performed. For functional training, lateral hops and SEBT was performed. And at the end, for resistance training, theraband was used with normal ankle joint movement. There is a progress in focus between the five domains over the 3weeks, as described below: The domains S and M are present across the whole intervention. In week 1, the main focus is on the A domain, in week 2 on the R domain, and in week 3 on the T domain. During the 3-week intervention period, 3 training sessions was held per week each lasting approximately 45 - 60 min, including 10 min warm up.
  Interventions: Other: SMART TRAINING
- Group B: Warm up exercises with foot intensive rehabilitation(FIRE) (Active Comparator): The FIRE intervention was included the progressive balance training, ankle and hip strengthening, range of motion exercises and foot massage. Plantar massage consisted of two, 1-min plantar massages with a 1-min rest between sets. Four previously established exercises were target the IFMs including the short-foot, toe-spread-out, hallux extension, and lesser-toe extension.
  Interventions: Other: FIRE training

INTERVENTIONS:
Other: SMART TRAINING — Patients in Group A received SMART training intervention. For sensory stimulation planter massage was given, and it was applied to entire planter surface. Grade III anterior to posterior talocrural joint mobilization was given (26). For balance, single and double leg stance was performed. For functional training, lateral hops and SEBT was performed. And at the end, for resistance training, theraband was used with normal ankle joint movement. There is a progress in focus between the five domains over the 3weeks, as described below: The domains S and M are present across the whole intervention. In week 1, the main focus is on the A domain, in week 2 on the R domain, and in week 3 on the T domain. During the 3-week intervention period, 3 training sessions was held per week each lasting approximately 45 - 60 min, including 10 min warm up
  Arms: Group A: warm up exercises with SMART training
Other: FIRE training — Patients in Group B was received foot intensive rehabilitation (FIRE).The FIRE intervention was include the progressive balance training, ankle and hip strengthening, range of motion exercises and foot massage. Plantar massage consisted of two, 1-min plantar massages with a 1-min rest between sets. Four previously established exercises were targeted the IFMs including the short-foot, toe-spread-out, hallux extension, and lesser-toe extension
  Arms: Group B: Warm up exercises with foot intensive rehabilitation(FIRE)

SUMMARY:
The study was a randomized clinical trial with the sample size of 26. The study was conducted at Sports Club Sheikhupura. Subjects were enrolled according to eligibility criteria. Patients were divided into two groups, each with 13 patients. Group A received SMART training intervention and warm-up exercises, while group B received Foot intensive rehabilitation exercises (FIRE) and warm up exercises. The session was around 45 to 60 min on each patient with three sessions per week on alternate days. A total of Three weeks treatment regime was given to the patients and assessment of patient's strength (CAIT) and performance (FAAM) was done at the baseline, after the completion of treatment at three weeks and after six weeks to observe the long-term effects.

DETAILED DESCRIPTION:
Ankle sprain is one of the most common sports injuries in physically active individuals and causes a high financial burden on the healthcare system. Seventy-four percent of patients with an acute ankle sprain suffered from residual symptoms lasting 29 months after the initial ankle sprain, such as pain, perceived instability, weakness and swelling. Lateral ankle sprains (LASs) are a common injury sustained by individuals who participate in recreational physical activities and sports. After LAS, a large proportion of individuals develop long-term symptoms, which contribute to the development of chronic ankle instability (CAI).The aim of this study to determine the comparative effects of SMART training intervention versus foot intensive rehabilitation (FIRE) on strength and performance in athletes with chronic ankle instability.

The study was a randomized clinical trial with the sample size of 26. The study was conducted at Sports Club Sheikhupura. Subjects was enrolled according to eligibility criteria. Patients was divided into two groups, each with 13 patients. Group A received SMART training intervention and warm-up exercises, while group B received Foot intensive rehabilitation exercises (FIRE) and warm up exercises. The session was around 45 to 60 min on each patient with three sessions per week on alternate days. A total of Three weeks treatment regime was given to the patients and assessment of patient's strength (CAIT) and performance (FAAM) was done at the baseline, after the completion of treatment at three weeks and after six weeks to observe the long-term effects.

ELIGIBILITY:
Inclusion Criteria:

* Athletes 18-45 years of age,
* 2 repeated episodes of giving way, feelings of instability
* Core training not less than 4 week.
* Chronic ankle instability more than 6 months.
* Repeated ankle sprain more than twice and patients with <24 points based on CAIT.
* Athletes with single side ankle instability

Exclusion Criteria:

* Acute concomitant injuries of the ankle.
* Individuals who were able to return to pre-injury levels of activity
* Serious lower-extremity injuries of the last 6 months
* Lower-extremity surgery, and neurological diseases
* Simultaneous severe sprain of both ankle joints

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Cumberland Ankle Instability Tool (CAIT) | Change from Baseline at 3 weeks and 6 weeks
  Cumberland Ankle Instability Tool (CAIT) was originally developed in English and proved to be of high content validity and good reliability. The main advantage of the questionnaire is that it consists of only 9 items, minimizing patient burden and increasing reliability. The precision of the instrument is increased as it is a multiple answer option instrument
Foot and Ankle Ability Measurement (FAAM) | Change from Baseline at 3 weeks and 6 weeks
  The Foot and Ankle Ability Measure (FAAM) assess the functional limitation of the foot and ankle. The FAAM has 29 items, scored between 0 and 4, divided into two sub-scales: activities of daily living (21 items) and sports (8 items)(24).For score analysis, the percentage of each sub scale is used separately. For FAAM ADL, person reliability is 0.87 and item reliability is0.99. For FAAM Sport, person reliability is 0.89 and item reliability is 1.0

CONTACTS AND LOCATIONS:
Overall Officials: wajeeha konain, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Sports Club Sheikhupura, Sheikhupura, Punjab Province, Pakistan

REFERENCES:
- [Background] Lin CI, Houtenbos S, Lu YH, Mayer F, Wippert PM. The epidemiology of chronic ankle instability with perceived ankle instability- a systematic review. J Foot Ankle Res. 2021 May 28;14(1):41. doi: 10.1186/s13047-021-00480-w. PMID 34049565
- [Background] Herzog MM, Kerr ZY, Marshall SW, Wikstrom EA. Epidemiology of Ankle Sprains and Chronic Ankle Instability. J Athl Train. 2019 Jun;54(6):603-610. doi: 10.4085/1062-6050-447-17. Epub 2019 May 28. PMID 31135209
- [Background] Al-Mohrej OA, Al-Kenani NS. Chronic ankle instability: Current perspectives. Avicenna J Med. 2016 Oct-Dec;6(4):103-108. doi: 10.4103/2231-0770.191446. PMID 27843798
- [Background] Abadi FH, Sankaravel M, Zainuddin FF, Elumalai G, Razli AI. The effect of aquatic exercise program on low-back pain disability in obese women. J Exerc Rehabil. 2019 Dec 31;15(6):855-860. doi: 10.12965/jer.1938688.344. eCollection 2019 Dec. PMID 31938709
- [Background] Delahunt E, Remus A. Risk Factors for Lateral Ankle Sprains and Chronic Ankle Instability. J Athl Train. 2019 Jun;54(6):611-616. doi: 10.4085/1062-6050-44-18. Epub 2019 Jun 4. PMID 31161942
- [Background] Hall EA, Chomistek AK, Kingma JJ, Docherty CL. Balance- and Strength-Training Protocols to Improve Chronic Ankle Instability Deficits, Part II: Assessing Patient-Reported Outcome Measures. J Athl Train. 2018 Jun;53(6):578-583. doi: 10.4085/1062-6050-387-16. Epub 2018 Jul 11. PMID 29995462
- [Background] Jaber H, Lohman E, Daher N, Bains G, Nagaraj A, Mayekar P, Shanbhag M, Alameri M. Neuromuscular control of ankle and hip during performance of the star excursion balance test in subjects with and without chronic ankle instability. PLoS One. 2018 Aug 13;13(8):e0201479. doi: 10.1371/journal.pone.0201479. eCollection 2018. PMID 30102713
- [Background] Kim J, Kang S, Kim SJ. A smart insole system capable of identifying proper heel raise posture for chronic ankle instability rehabilitation. Sci Rep. 2022 Jun 24;12(1):10796. doi: 10.1038/s41598-022-14313-8. PMID 35750787
- [Background] Molla-Casanova S, Ingles M, Serra-Ano P. Effects of balance training on functionality, ankle instability, and dynamic balance outcomes in people with chronic ankle instability: Systematic review and meta-analysis. Clin Rehabil. 2021 Dec;35(12):1694-1709. doi: 10.1177/02692155211022009. Epub 2021 May 31. PMID 34058832